CLINICAL TRIAL: NCT02353806
Title: Pharmacokinetics of Amlodipine Besylate at Delivery and During Lactation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jamie Morgan, Maternal Fetal Medicine Fellow, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042014-059; UL1TR001105 (NIH)
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hypertension in Pregnancy
Keywords: Amlodipine besylate; Breast milk; Pharmacokinetics; Chronic hypertension; Pregnancy
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women taking amlodipine (Experimental): Women already taking amlodipine besylate 5 mg for treatment of chronic hypertension in pregnancy who plan to breastfeed postpartum will be assigned to the single experimental arm.
  Interventions: Drug: Amlodipine besylate

INTERVENTIONS:
Drug: Amlodipine besylate — Pregnant and postpartum women will continue taking amlodipine besylate 5 mg for treatment of chronic hypertension as prescribed by their clinician.

SUMMARY:
This is a phase IV prospective trial to collect and analyze information about the maternal pharmacokinetics of amlodipine besylate at the time of delivery and during postpartum lactation. The study will also evaluate amlodipine concentrations in the infants of breastfeeding mothers who are taking amlodipine besylate for treatment chronic hypertension.

DETAILED DESCRIPTION:
We plan to evaluate the pharmacokinetics of amlodipine besylate at the time of delivery, to determine if transplacental passage of the drug occurs. We will also examine the drug kinetics in postpartum lactation to establish whether amlodipine is excreted into breast milk. The outcomes of interest are plasma concentration of amlodipine at delivery and the drug concentrations in blood and breast milk over a twenty-hour steady-state period following milk-supply establishment. Fifteen patients already taking 5 mg of amlodipine during pregnancy for the treatment of chronic hypertension will be recruited from the antepartum Obstetric Complications Clinic at Parkland Hospital. Only women who are breastfeeding will be eligible for the study. Patients who elect to participate in the study will continue their amlodipine 5 mg dosing through delivery and into the postpartum period. Maternal blood will be drawn within one hour of delivery and fetal cord blood collected at the time of delivery. Patients will then have blood drawn over a 24 hour period beginning on postpartum day 2 after delivery following administration of their once-daily amlodipine dose. At each blood draw, the patient will also use a breast pump to express breast milk for paired analysis. Both blood and breast milk amlodipine levels will be calculated for all samples. The levels will be used to determine the pharmacokinetics of amlodipine in the peri- and postpartum patient, including concentrations in plasma and breast milk.

In addition to collecting maternal data, a range of clinical information will be collected on each study patient's infant including weight, Apgar scores, hemodynamic parameters, physical examination and hospital course. This information will be used to screen for any potential complications associated with infant exposure to amlodipine. An infant blood sample will also be obtained in conjunction with the routine neonatal blood collection that occurs at 1-2 days of postnatal life and this will be analyzed to determine serum amlodipine concentration in breastfeeding infants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Pregnant female
* Already taking amlodipine 5 mg for treatment of chronic hypertension in pregnancy;
* Hospitalized following routine term vaginal delivery or uncomplicated cesarean delivery
* Breastfeeding or breast and bottle-feeding their infant

Exclusion Criteria:

* Known kidney disease
* Delivery complicated by chorioamnionitis, endometritis or postpartum hemorrhage
* Administration of greater than 5 mg of amlodipine in 24 hour period

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Morgan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant Women Taking Amlodipine
Started | 16
Completed | 6
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | NA — This study only included pregnant women.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  Hispanic | 12
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Amlodipine in the Maternal Serum
Description: The time to peak amlodipine concentration in the maternal serum in the peripartum period was be measured.
Time Frame: Maternal blood samples will be obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Population: Although 16 women were enrolled in the study, only 11 of the 16 had blood drawn at the time of delivery. This was due to limitations of study personnel availability to attend the deliveries of all study patients
Measure: Mean (Standard Deviation); unit: (hr*ng)/mL
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
(hr*ng)/mL | 53.4 (19.8)

2. Primary Outcome: Time to Maximal Concentration in the Maternal Serum.
Description: The time to reach maximal amlodipine concentration in the maternal serum in the peripartum period was measured.
Time Frame: Maternal blood samples were obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Population: Although 16 women were enrolled in the trial, only 11 had their blood drawn at the time of delivery due to limited availability of study personnel.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
Hours | 7.5 (1.5)

3. Primary Outcome: Maximal Amlodipine Maternal Serum Concentration
Description: The maximum concentration of amlodipine detected in the maternal serum in the peripartum period was measured.
Time Frame: Maternal blood samples were obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
ng/mL | 2.0 (1.0)

4. Primary Outcome: Half-life of Amlodipine in Maternal Plasma
Description: The half-life of amlodipine in the maternal plasma in the peripartum period was measured.
Time Frame: Maternal blood samples were obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
Hours | 13.7 (4.9)

5. Primary Outcome: Clearance Rate of Plasma Amlodipine
Description: The clearance rate of amlodipine from the maternal plasma was measured.
Time Frame: Maternal blood samples were obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
L/hr | 109.7 (58.9)

6. Primary Outcome: Drug Levels/Concentration in Cord Blood (Amlodipine Levels/Concentrations)
Description: Maternal and cord blood amlodipine levels/concentrations will be determined.
Time Frame: Pair maternal blood sample and cord blood sample will draw within 1 hour of delivery
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 11
ng/mL
  Infant cord blood plasma amlodipine concentration | 0.49 (0.29)
  Maternal serum amlodipine concentration | 1.27 (0.84)

7. Primary Outcome: Amlodipine Concentration in Breastmilk
Description: The concentration of amlodipine besylate was measured in breastmilk samples.
Time Frame: Breast milk samples were obtained at 4, 6, 8, 12, 15 and 24 hours after amlodipine dosing
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 6
ng/mL | NA (NA) — Amlodipine concentrations in maternal breast milk were undetectable at the lower limit of assay detection (<0.1 ng/mL).

8. Primary Outcome: Drug Level/Concentration in Infant Blood (Amlodipine Level/Concentration)
Description: Infant amlodipine level/concentration will be determined.
Time Frame: Infant blood sample drawn at approximately 36 hours of life
Population: Of the 16 patients enrolled in the study, only 8 continued in the study and allowed their infant's to have study sampling performed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pregnant Women Taking Amlodipine
Number analyzed (Participants) | 8
ng/mL | NA (NA) — Amlodipine concentrations in infant plasma were undetectable at the lower limit of assay detection (<0.1 ng/mL)

9. Secondary Outcome: Neonatal Birth Weight
Description: The neonatal weight at birth was collected.
Time Frame: Neonatal weight at the time of birth.
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Infant's Born to Women Taking Amlodipine Besylate: Infant's born to women already taking amlodipine besylate 5 mg for the treatment of chronic hypertension in pregnancy and who planned to breastfeed their babies.
  Amlodipine besylate: Pregnant and postpartum women will continue taking amlodipine besylate 5 mg for treatment of chronic hypertension as prescribed by their clinician.
Arm/Group | Infant's Born to Women Taking Amlodipine Besylate
Number analyzed (Participants) | 16
grams | 3281 (525)

10. Secondary Outcome: Infant Gestational Age at Delivery.
Description: The mean gestational age of infants born to mothers taking Amlodipine besylate 5 mg daily was collected.
Time Frame: Gestational age at the time of birth
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Infant's Born to Women Taking Amlodipine Besylate: Infant's born to women already taking amlodipine besylate 5 mg for the treatment of chronic hypertension in pregnancy and who planned to breastfeed their babies.
Arm/Group | Infant's Born to Women Taking Amlodipine Besylate
Number analyzed (Participants) | 16
weeks | 38.2 (0.8)

11. Secondary Outcome: Infant Length of Stay.
Description: The length of stay of infants born to women taking amlodipine besylate will be collected.
Time Frame: Time from birth to hospital discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Infant's Born to Women Taking Amlodipine Besylate
Number analyzed (Participants) | 16
Days | 3.6 (0.5)

12. Secondary Outcome: Major Infant Complications
Description: Any major complications experienced by infants born to women taking amlodipine besylate including NICU admission, intraventricular hemorrhage, neonatal seizures, need for respiratory support and apnea were collected.
Time Frame: During neonatal hospitalization
Measure: Number; unit: Participants
Arm/Group | Infant's Born to Women Taking Amlodipine Besylate
Number analyzed (Participants) | 16
Participants
  Admission to the NICU | 0
  Major neonatal complications (IVH, apnea, seizure) | 0

ADVERSE EVENTS:
Arm/Group | Pregnant Women Taking Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No